CLINICAL TRIAL: NCT06601738
Title: Effects Of Isometrics and Dynamic Handgrip Exercise Training On Cardiovascular Parameters In Hypertensive Patients
Brief Title: Isometric and Dynamic Handgrip Training Effects on Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Arisha Noor
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Hypertension
Keywords: Systolic Blood Pressure; Diastolic Blood Pressure; Mean Arterial Blood Pressure; Pulse Pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental)
  Interventions: Other: Isomeric Hand Grip Exercises
- Group B (Active Comparator)
  Interventions: Other: Dynamic Hand Grip Exercises

INTERVENTIONS:
Other: Isomeric Hand Grip Exercises — Patients will be instructed to squeeze and sustain the dynamometer for 2 min at 30% M.V.C. The dynamometer pointer which read the scale provided visual feedback to the subjects for the maintenance of the 30% M.V.C. This procedure will be repeated twice for each training session with a 5-minute rest in between.
  Arms: Group A
Other: Dynamic Hand Grip Exercises — Dynamic handgrip exercise was performed with both-sided, metronome-guided rhythmic hand contractions for 2min. The handgrip ring, closest to 20% of MVC, was chosen for DHE which was performed at a frequency of 30/min, acoustically indicated by a metronome beat.
  Arms: Group B

SUMMARY:
Essential hypertension accounts for 13 percent of total deaths worldwide, accounting for one of the major risk factors. Hypertension (high blood pressure) is when the pressure in your blood vessels is too high (140/90 mmHg or higher). Dynamic exercises, sustained hand grip contractions elicit lower systolic blood pressure and heart rate responses. So for patients undergoing exercise therapy, low intensity isometric exercises are preferable. Significant reduction is seen in mean arterial blood pressure and systolic blood pressure in individuals conducting isometric for 8 weeks in 30%. The reduction in systolic blood pressure will be clinically significant. The main objective of this study will be to determine the effects of dynamic and isometric handgrip exercise training on cardiovascular parameters in hypertensive patients Grade 1 hypertensive patients are included as per AHA and JNC7 criteria. A sample of 100 hypertensive patients will be recruited and divided into two treatment groups; G1: dynamic exercise in hypertensive patients, and G2: isometric exercise in hypertensive patients. Outcome measure will include systolic blood pressure, diastolic blood pressure, mean arterial blood pressure and pulse pressure. Outcome measures will be assessed at baseline and 2nd and 4th weeks posttreatment.

DETAILED DESCRIPTION:
Hypertension is one of the most prevalent diseases leading to morbidity and mortality, affecting millions of people every year. Pharmaceutical management is the main treatment method used. Exercise therapy mainly isometrics and dynamic handgrip exercises provide a non pharmacological management leading to decrease in symptoms. The association of hypertension with physical inactivity, sedentary behavior, and occupational exposure to chemicals, obesity, older age, genetics, being overweight or obese, not being physically active, ,high-salt diet, job insecurity, job loss, and the psychosocial work environment and drinking too much alcohol. Lifestyle changes like eating a healthier diet, quitting tobacco, and being more active can help lower blood pressure. Hypertension rates are strongly associated with age. Acute effects of isometric and dynamic handgrip exercise on cardiovascular parameters in hypertensive subjects are numerous . They may also have some adverse effects on the cardiorespiratory system, particularly, through the elevation of blood pressure.

Since an acute bout of exercise can transiently improve cardiovascular endothelial function, arterial stiffness, and ambulatory blood pressure. The dynamic handgrip exercise is performed by repetitive contraction and relaxation of the hand at a maximum frequency. In order to determine the intensity of handgrip exercises, maximum isometric handgrip strength of the right and left hand was measured with a handgrip dynamometer. Isometric exercises differ from dynamic exercises because in this there is no change in muscle length or static force. Single handgrip exercise could reduce the blood pressure for couple of hours so a patient can perform this exercise several times a day if not being fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Gender (both)
* Age (30-55 years)
* Grade 1 hypertensive patients as per AHA and JNC7 criteria

Exclusion Criteria:

* Patients having hypertension associated due to other diseases.
* Patients having joint problems of wrist, hand fingers, ligament and tendon injuries of hand and fingers.
* Patients having recent hand surgeries, fracture, history of arthritis, carpal tunnel syndrome.
* Patient having history of any symptoms of chest pain.
* Patients having loss of consciousness during physical activity.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-08-30 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
6 Minute Walk test | Baseline; 4nd Week; 8th Week
  It is a standard method for measuring exercise capacity in patients with cardiopulmonary disease such as PAH. The 6MWT measures how far a patient can walk in 6 minutes. Walking is an activity performed every day by most patients except for those most severely limited. By assessing patients' ability to exercise, the 6MWT provides a global assessment of respiratory, cardiovascular, neuromuscular, and cognitive function. The 6MWT does not differentiate what limits the patient nor does it assess maximal exercise capacity. Instead, the 6MWT allows the patient to exercise at a daily functional level and is a useful tool for assessing severity of disease, and increasing walk distance correlates with a subjective improvement in dyspnea
Blood Pressure Measurements (SBP & DBP) | Baseline; 4nd Week; 8th Week
  An appropriately sized cuff for the arm circumference was installed on the non-dominant arm. Blood pressure was measured every 20 minutes by 24 hours, and awake and sleep periods were determined according to information provided by the patients, the following are 7 strategies recommended by the AHA/AMA for accurate attainment of BP: 1) no conversation, 2) empty bladder, 3) use correct cuff size, 4) place BP cuff on bare arm, 5) support arm at heart level, 6) keep legs uncrossed, and 7) support back and feet

CONTACTS AND LOCATIONS:
Overall Officials: Arisha Noor, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehabiliation Clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oliveira-Silva L, Fecchio RY, Silva Junior NDD, Pio-Abreu A, Silva GVD, Drager LF, Silva de Sousa JC, Forjaz CLM. Post-dynamic, isometric and combined resistance exercise responses in medicated hypertensive men. J Hum Hypertens. 2024 Jan;38(1):52-61. doi: 10.1038/s41371-023-00859-1. Epub 2023 Sep 5. PMID 37670145
- [Background] Ogbutor GU, Nwangwa EK, Uyagu DD. Isometric handgrip exercise training attenuates blood pressure in prehypertensive subjects at 30% maximum voluntary contraction. Niger J Clin Pract. 2019 Dec;22(12):1765-1771. doi: 10.4103/njcp.njcp_240_18. PMID 31793486
- [Background] Cahu Rodrigues SL, Farah BQ, Silva G, Correia M, Pedrosa R, Vianna L, Ritti-Dias RM. Vascular effects of isometric handgrip training in hypertensives. Clin Exp Hypertens. 2020;42(1):24-30. doi: 10.1080/10641963.2018.1557683. Epub 2019 Jan 9. PMID 30626217
- [Background] Punia S, Kulandaivelan S. Home-based isometric handgrip training on RBP in hypertensive adults-Partial preliminary findings from RCT. Physiother Res Int. 2020 Jan;25(1):e1806. doi: 10.1002/pri.1806. Epub 2019 Aug 16. PMID 31418966
- [Background] Polito MD, Papst R, Goessler K. Twelve weeks of resistance training performed with different number of sets: Effects on maximal strength and resting blood pressure of individuals with hypertension. Clin Exp Hypertens. 2021 Feb 17;43(2):164-168. doi: 10.1080/10641963.2020.1833024. Epub 2020 Oct 10. PMID 33043697
- [Background] Kappus RM, Bunsawat K, Brown MD, Phillips SA, Haus JM, Baynard T, Fernhall B. Effect of oxidative stress on racial differences in vascular function at rest and during hand grip exercise. J Hypertens. 2017 Oct;35(10):2006-2015. doi: 10.1097/HJH.0000000000001433. PMID 28594709
- [Background] Fecchio RY, de Sousa JCS, Oliveira-Silva L, da Silva Junior ND, Pio-Abreu A, da Silva GV, Drager LF, Low DA, Forjaz CLM. Effects of dynamic, isometric and combined resistance training on blood pressure and its mechanisms in hypertensive men. Hypertens Res. 2023 Apr;46(4):1031-1043. doi: 10.1038/s41440-023-01202-4. Epub 2023 Feb 9. PMID 36759659